CLINICAL TRIAL: NCT06667908
Title: A Phase 2, Randomized, Open-Label, Active-Controlled Study of JNJ-90301900 in Combination With Chemoradiation Followed by Durvalumab in Locally Advanced and Unresectable Stage III NSCLC
Brief Title: A Study of JNJ-90301900 in Combination With Chemoradiation Followed by Consolidation Immunotherapy for Non-Small Cell Lung Cancer (NSCLC)
Acronym: CONVERGE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Enterprise Innovation Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90301900NSC2001; 90301900NSC2001 (Other: Janssen Research & Development, LLC); 2024-518276-32-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Cohort A and Cohort B (Experimental): Participants will receive JNJ-90301900 injected intratumorally and/or intranodally (cohort A: 22% gross tumor volume [GTV] and cohort B: 33% GTV) along with cCRT (concurrent chemotherapy with radiation therapy) followed by consolidation immunotherapy (cIT) to evaluate feasibility of JNJ-90301900 injection procedure.
  Interventions: Drug: JNJ-90301900; Biological: Durvalumab; Radiation: Concurrent Chemo/Radiation Therapy (cCRT); Drug: Concurrent Chemo/Radiation Therapy (cCRT): Carboplatin; Drug: Concurrent Chemo/Radiation Therapy (cCRT): Paclitaxel
- Part 2: Arm A and Arm B (Experimental): Participants will receive JNJ-90301900 injected intratumorally and/or intranodally (Arm A: 22% GTV and Arm B: 33% GTV) along with cCRT followed by cIT to evaluate the efficacy and safety of JNJ-90301900.
  Interventions: Drug: JNJ-90301900; Biological: Durvalumab; Radiation: Concurrent Chemo/Radiation Therapy (cCRT); Drug: Concurrent Chemo/Radiation Therapy (cCRT): Carboplatin; Drug: Concurrent Chemo/Radiation Therapy (cCRT): Paclitaxel
- Part 2: Arm C: (Control treatment) (Active Comparator): Participants will receive treatment with cCRT followed by cIT as control treatment to evaluate the efficacy and safety of JNJ-90301900.
  Interventions: Biological: Durvalumab; Radiation: Concurrent Chemo/Radiation Therapy (cCRT); Drug: Concurrent Chemo/Radiation Therapy (cCRT): Carboplatin; Drug: Concurrent Chemo/Radiation Therapy (cCRT): Paclitaxel

INTERVENTIONS:
Drug: JNJ-90301900 — JNJ-90301900 will be injected intratumorally and/or intranodally.
  Arms: Part 1: Cohort A and Cohort B; Part 2: Arm A and Arm B
Biological: Durvalumab — Durvalumab will be administered as intravenous (IV) infusion as cIT.
Radiation: Concurrent Chemo/Radiation Therapy (cCRT) — Radiation by intensity modulated radiation therapy (IMRT) will be administered.
Drug: Concurrent Chemo/Radiation Therapy (cCRT): Carboplatin — Carboplatin will be administered as IV infusion as platinum-based doublet chemotherapy.
Drug: Concurrent Chemo/Radiation Therapy (cCRT): Paclitaxel — Paclitaxel will be administered as IV infusion as platinum-based doublet chemotherapy.

SUMMARY:
The purpose of this study is to determine whether JNJ-90301900 added to concurrent platinum-based doublet chemotherapy with radiation therapy (cCRT) followed by consolidation immunotherapy (cIT) can improve objective response rate (ORR; that is percentage of participants whose best response is complete response or partial response during the study) in participants with locally advanced and unresectable stage III non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must be a candidate for standard of care (SOC) treatment of non small cell lung cancer (NSCLC) by concurrent platinum-based doublet chemotherapy with radiation therapy (cCRT) followed by consolidation durvalumab treatment as determined by the investigator and per local guidelines at screening
* Have a medical history of pathologically (histologically or cytologically) proven diagnosis of NSCLC within 3 months prior to enrollment/randomization
* Have locally advanced unresectable stage III NSCLC according to the eighth edition lung cancer stage classification
* Have at least 1 target lesion (primary lung lesion or involved lymph node[s]) per RECIST version 1.1 that is amenable to intratumoral and/or intranodal injection and intensity modulated radiation therapy (IMRT) as determined by the investigator at screening
* Have an eastern cooperative oncology group (ECOG) performance status of 0 to 1

Exclusion Criteria:

* Medical history of: (a) Primary immunodeficiency (b) Organ transplant that requires therapeutic immunosuppression
* Any of the following within 3 months prior to enrollment/randomization: severe or unstable angina, myocardial infarction, clinically significant ventricular arrhythmias or heart failure New York heart association functional classification class III to IV
* Another concurrent or prior primary malignancy within the last 36 months at informed consent
* Known allergies, hypersensitivity, or intolerance to any ingredients of JNJ-90301900 crystalline solution, platinum-based doublet chemotherapy (ChT), or durvalumab
* History of coagulation disorders, including: (a) Active bleeding diathesis or requirement for therapeutic anticoagulation or antiplatelet that cannot be interrupted or altered for JNJ-90301900 injection procedures, (b) Major thromboembolic events (for example, pulmonary embolism, cerebrovascular accident) within 3 months of enrollment or randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Using Independent Central Review (ICR) Assessment | Up to 2 Years and 2 months
  ORR is defined as the percentage of participants who have a best response of complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors (RECIST) version (v) 1.1 using ICR assessments.

SECONDARY OUTCOMES:
Disease Response Rate (ORR) Post-cCRT and Pre-cIT | Up to 12 Weeks
  Disease response rate is defined as percentage of participants who achieve CR or PR, post-concurrent platinum-based doublet chemotherapy with radiation therapy (cCRT) and pre-consolidation immunotherapy (cIT) based on investigator's assessment according to RECIST v1.1.
Disease Control Rate (DCR) Post-cCRT and Pre-cIT | Up to 12 Weeks
  DCR is defined as percentage of participants who achieve CR, PR and stable disease post-cCRT and pre-cIT based on investigator's assessment according to RECIST v1.1.
Objective Response Rate (ORR) as Assessed by the Investigator | Up to 2 Years and 2 months
  ORR is defined as the percentage of participants who have a best response of CR or PR using RECIST v1.1 as assessed by the investigator.
Progression Free Survival (PFS) | Up to 2 Years and 2 months
  PFS is defined as the time from the enrollment/randomization until disease progression or death due to any cause according to RECIST v1.1.
Duration of Response (DoR) | Up to 2 Years and 2 months
  DoR will be calculated among responders from the date of initial documentation of a response to the date of first documented evidence of relapse according to RECIST v1.1, or death due to any cause, whichever occurs first.
Time to Locoregional Failure (LRF) | Up to 2 Years and 2 months
  Time to LRF is defined as the time from enrollment/randomization to the first LRF using ICR assessments.
Time to Distant Failure (DF) | Up to 2 Years and 2 months
  Time to DF is defined as the time from enrollment/randomization to the first DF using ICR assessments.
Number of Participants with Treatment-Emergent Adverse Event (TEAE) Related to Study Treatment | Up to 2 Years and 2 months
  TEAE is defined as any new or worsening adverse event (AE) occurring at or after the initial administration of study treatment through the day of last dose of study treatment received plus 30 days or prior to the start of subsequent anticancer therapy (non-durvalumab), whichever is earlier, or any follow-up AE with onset date and time beyond 30 days after the last dose of study treatment but prior to the start of subsequent anticancer therapy, or any AE that is considered treatment-related regardless of the start date of the event. TEAEs related to JNJ-90301900 injection procedure, JNJ-90301900, RT, ChT, or cIT will be reported.
Number of Participants Reporting Laboratory Parameters, Physical Examination, Vital Signs Including Eastern Cooperative Oncology Group (ECOG) Performance Status Abnormalities | Up to 2 Years and 2 months
  Participants with laboratory parameters, physical examination, vital signs including ECOG performance status abnormalities will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Enterprise Innovation Inc. Clinical Trial, Study Director — Johnson & Johnson Enterprise Innovation Inc.
Locations (33):
- United States (12):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - Orlando Health Cancer Institute, Orlando, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - FirstHealth of the Carolinas, Pinehurst, North Carolina
  - Oregon Health And Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
- Australia (3):
  - Sir Charles Gairdner Hospital, Nedlands
  - Macquarie University, North Ryde
  - Royal Melbourne Hospital, Parkville
- Brazil (3):
  - Fundacao Pio XII, Barretos
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- France (5):
  - Hopital De La Cavale Blanche, Brest
  - Hopital Nord Marseille, Marseille
  - Hopital Tenon, Paris
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Prince of Wales Hospital, Shatin, Hong Kong
- Netherlands (2):
  - Antoni van Leeuwenhoek, Amsterdam
  - Radboud Umcn, Nijmegen
- Spain (4):
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Univ. I Politecni La Fe, Valencia
- Turkey (Türkiye) (2):
  - Marmara University Pendik Training Hospital, Istanbul
  - Sakarya University Training and Research Hospital, Sakarya
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency